CLINICAL TRIAL: NCT05091671
Title: Investigating the Effectiveness of the "Free From Pain" Exercise and Education Programme in Decreasing Early Osteoarthritic / Generalised Musculoskeletal Pain in People Over 60 Years of Age
Brief Title: Free From Pain Exercise Programme Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Talita Cumi Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FFPETFETS004
Record Dates: First submitted 2021-10-12; First posted 2021-10-25 (Actual); Last update posted 2022-10-21 (Actual); Status verified 2022-10

CONDITIONS: Musculoskeletal Pain; Fear of Falling
MeSH Terms: conditions — Musculoskeletal Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Free From Pain Exercise Programme Variation 1 (Active Comparator): Participants will have the initial online consultation and will be provided with the exercise booklet and the 12 information/metaphor leaflets. The ongoing 12 Zoom online sessions are not included in this option. Instead, participants will be asked to independently engage in the exercises within the exercise booklet. They will be advised to either do all 3 sets of exercises 3 times a week or to do the neck and low back exercises twice a week and the Otago exercises 3 times a week. The exercises should take around an hour to complete each day. The ideal plan would be as follows:
  Monday - Otago exercises. Tuesday - Neck and Back exercises. Wednesday - Otago exercises. Thursday - Rest day. Friday - Neck and Back exercises. Saturday - Otago exercises. Sunday - Rest day.
  Interventions: Other: Free From Pain Exercise Programme Variation 1
- Free From Pain Exercise Programme Variation 2 (Experimental): Participants will have the initial online consultation and will be provided with the exercise booklet and12 information/metaphor leaflets. This variation also includes the online zoom sessions. The online zoom session will involve a short presentation and a group discussion for 15 minutes followed by a 45-minute exercise class which will be delivered by a suitably trained individual. The exercise class will include the exercises from the Otago Exercise programme + the Motor Control Exercises for low back pain + Isometric and strengthening exercise for the neck. Participants assigned to this intervention will also be asked to independently engage in the exercises within the exercise booklet. They will be advised to use the same weekly structure described previously.
  Interventions: Other: Free From Pain Exercise Programme Variation 2

INTERVENTIONS:
Other: Free From Pain Exercise Programme Variation 1 — Includes the initial 45-minute consultation + the exercise booklet + the 12 reasons to exercise leaflets + the 12 metaphor leaflets.
  Arms: Free From Pain Exercise Programme Variation 1
Other: Free From Pain Exercise Programme Variation 2 — Includes the initial 45-minute consultation + the exercise booklet + the 12 reasons to exercise leaflets + the 12 metaphor leaflets, and the 12 Zoom online sessions.
  Arms: Free From Pain Exercise Programme Variation 2

SUMMARY:
To determine the effectiveness of the "Free from Pain" exercise and information programme. The complete programme provides exercises and information for people over the age of 60 to reduce early osteoarthritic and generalised musculoskeletal pain and fear of falling. The study will compare the effects of 2 versions of the Free from Pain programme to ascertain which is the most effective.

DETAILED DESCRIPTION:
Chronic musculoskeletal conditions are the leading cause of disability worldwide. The World Health Organization estimates that approximately 1.71 billion people have musculoskeletal conditions worldwide. They cause a significant economic burden on the NHS. £5 billion of England's yearly NHS budget goes towards the treatment of musculoskeletal conditions.

Disability from the initial pain is worsened by immobility, which will cause a loss of muscle mass and fitness and an increased risk of falls, further injury, and diseases associated with poor activity (such as heart attacks and some cancers). In chronic musculoskeletal pain conditions, providing information and participating in exercise programmes are commonly used. However, there are no evidence-based recommendations on which plans are the most effective.

The "Free from Pain" exercise programme is a fusion of three different generally accepted exercise programmes. Therapeutic exercise programmes exist for individual body parts, but there is no single generalised exercise programme that targets all body parts. Hence, the creation of this fusion of programmes. The three programmes are the Otago exercises for lower body strength and balance, the motor control exercises for the lower back and the isometric exercises for the neck and shoulder. The Otago exercise program (OEP) was developed by Robertson and Campbell for the New Zealand accident compensation corporation (ACC). The aim of the programme was to improve balance and strength in patients to prevent falls. The Otago exercise programme has also been identified as an effective intervention in community-dwelling older adults for coping with musculoskeletal pain.

Educational information leaflets will also be provided as part of the programme. These comprise an introductory leaflet, in addition to 12 reasons to exercise and 12 metaphor leaflets. The 12 reasons to exercise leaflets provide evidence-based information regarding the effects exercise can have on health. The 12 metaphor leaflets will contain metaphors used by the lead investigator in his practice over many years. These metaphors attempt to link everyday life with health, allowing laypersons to better understand the importance of certain lifestyle choices in regard to maintaining health. It will be recommended to participants that they read one reason to exercise leaflet and one metaphor each week for 12 weeks to ensure that they absorb the information fully and do not overbear themselves with information.

This is a randomised control trial feasibility study which will be conducted over an 18-month period, during which participants will be asked to provide data in the form of completed surveys three times, at baseline, 3 months, and 6 months. The aim of this randomised control trial feasibility study is to determine the effectiveness of the "Free from Pain" exercise and information programme. The complete programme provides exercises and information for people over the age of 60 in reducing early osteoarthritic and generalised musculoskeletal pain and fear of falling. The study will compare the effects of 2 versions of the Free from Pain programme to ascertain which is the most effective.

The study population will include 60 participants who will be split into 2 groups. One group will carry out the exercise classes independently at home, whereas the other group will participate in the online zoom exercise classes with a trained individual leading the class.

ELIGIBILITY:
Inclusion Criteria:

* 60 years of age +
* Has early osteoarthritic / generalised musculoskeletal pain

Exclusion Criteria:

* Lacking the physical ability or cardiovascular fitness required to participate in an exercise programme. This criterion will be explained on the participant information sheet by stating, "If you are unable to walk up a flight of stairs without getting breathless, please do not apply for participation in this study". This will also be confirmed in the initial consultation, during which Dr. Ampat will once again ask participants this question.
* Self-reported lack of mental ability to participate in the exercise programme.
* Have had a lower-limb joint (hip or knee) replacement, as some of the exercises may be contra-indicative to these conditions.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-02-28 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in Musculoskeletal Health Questionnaire scores (MSK-HQ) | Baseline, 3 weeks, 6 weeks, 3 months and 6 months
  Participants will be asked to report changes in Musculoskeletal Health Questionnaire scores to assess changes in musculoskeletal pain. The MSK-HQ is scored on a range of 0-56, with a higher score indicating better MSK-HQ health status.
Changes in Pain as assessed by a Visual Analogue Scale (VAS) | Baseline, 3 weeks, 6 weeks, 3 months and 6 months
  Changes in pain in the back, hips, knees, ankles and feet will be assessed via a self-report Visual Analogue Scale (VAS) as follows: 0 to 10 where 0 is 'No Pain' and 10 is 'The worst imaginable pain', with total scoring range of 0-50.

SECONDARY OUTCOMES:
Usefulness scale for patient information material (USE) | 6 months
  Reports using the usefulness scale for patient information material (USE) will be collected to assess the usefulness of the information leaflets provided. A maximum total score of 90 suggests that the participant 'completely agrees' with nine positive statements regarding the usefullness of the information material provided, whilst a minimum score of 0 suggests that they 'completely disagree' with said statements.
Changes in Short Falls Efficacy Scale International (Short FES-I) | Baseline, 3 weeks, 6 weeks, 3 months and 6 months
  Changes in scores on the Short Falls Efficacy Scale Internation (short FES-I) to assess improvements regarding fear of falling, where a minimum score of 7 means 'no concern about falling' and a maximum score of 28 means 'severe concern about falling'.
6-point Likert Scale | 6 months
  Upon completion of the study, participants will be asked to rate on a 0-5 likert scale (where 0 means 'extremely likely' and 5 means 'extremely unlikely') how likely they are to recommend the exercise programme to friends or family who may require it.

OTHER OUTCOMES:
Emergence of adverse effects in the form of additional pain as assessed by a Visual Analogue Scale (VAS). | 6 months
  Participants will be asked to refer to a 0-10 VAS pain scale (where 0 denotes pain-free and 10 denotes worst pain possible) if they experience any unexpected pain throughout the study period. If they experience pain which they determine to be 2 points higher on this scale than their pain level at the study onset, which they beleive to be as a result of the exercises, they will be asked to contact the research team, who will remove them from the study. The number of participants who are forced or wish to withdraw due to increased pain will be recorded and analysed to further ascertain the suitability and safety of the intervention.
Recruitment and retention rates as assessed by summary statistics and 95% confidence intervals. | 6 months
  Recruitment and retention rates will be reported using summary statistics and 95% confidence intervals to determine feasibility and sample size for the full trial.

CONTACTS AND LOCATIONS:
Overall Officials: George Ampat, Principal Investigator — National Health Service
Locations (1):
- Talita Cumi LTD., Southport, Merseyside, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
At the end of the study, data will be fully anonymised. Only non-identifiable, anonymised data will be archived along with the publication for use of other researchers. For instance, the age, sex, and study results of participants will be archived indefinitely as a supplementary document to the publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will become available at the completion of the study on 31/12/2022. It will be available for other researchers indefinitely.
Access Criteria: The non-identifiable data will be openly available as a supplementary document to the publication.

REFERENCES:
- [Background] Hill JC, Kang S, Benedetto E, Myers H, Blackburn S, Smith S, Dunn KM, Hay E, Rees J, Beard D, Glyn-Jones S, Barker K, Ellis B, Fitzpatrick R, Price A. Development and initial cohort validation of the Arthritis Research UK Musculoskeletal Health Questionnaire (MSK-HQ) for use across musculoskeletal care pathways. BMJ Open. 2016 Aug 5;6(8):e012331. doi: 10.1136/bmjopen-2016-012331. PMID 27496243
- [Background] Kempen GI, Yardley L, van Haastregt JC, Zijlstra GA, Beyer N, Hauer K, Todd C. The Short FES-I: a shortened version of the falls efficacy scale-international to assess fear of falling. Age Ageing. 2008 Jan;37(1):45-50. doi: 10.1093/ageing/afm157. Epub 2007 Nov 20. PMID 18032400
- [Background] Holzel LP, Ries Z, Dirmaier J, Zill JM, Kriston L, Klesse C, Harter M, Bermejo I. Usefulness scale for patient information material (USE) - development and psychometric properties. BMC Med Inform Decis Mak. 2015 Apr 19;15:34. doi: 10.1186/s12911-015-0153-7. PMID 25927192
- [Result] World Health Organisation (WHO) (2021). Musculoskeletal Conditions [Fact Sheet]. [Cited January 2021]. Retrieved from: https://www.who.int/news-room/fact-sheets/detail/musculoskeletal-conditions
- [Result] Arthritis Research UK. Understanding Arthritis: A Parliamentary Guide to Musculoskeletal Health. Chesterfield: Arthritis Research UK; 2013.
- [Result] Baker MK, Atlantis E, Fiatarone Singh MA. Multi-modal exercise programs for older adults. Age Ageing. 2007 Jul;36(4):375-81. doi: 10.1093/ageing/afm054. Epub 2007 May 30. PMID 17537741
- [Result] Gillespie LD, Robertson MC, Gillespie WJ, Sherrington C, Gates S, Clemson LM, Lamb SE. Interventions for preventing falls in older people living in the community. Cochrane Database Syst Rev. 2012 Sep 12;2012(9):CD007146. doi: 10.1002/14651858.CD007146.pub3. PMID 22972103
- [Result] Hedley L, Suckley N, Robinson L, Dawson P. Staying Steady: a community-based exercise initiative for falls prevention. Physiother Theory Pract. 2010 Oct;26(7):425-38. doi: 10.3109/09593980903585059. PMID 20673075
- [Result] Nyman SR, Victor CR. Older people's participation in and engagement with falls prevention interventions in community settings: an augment to the Cochrane systematic review. Age Ageing. 2012 Jan;41(1):16-23. doi: 10.1093/ageing/afr103. Epub 2011 Aug 28. PMID 21875865
- [Result] Stiggelbout M, Hopman-Rock M, Crone M, Lechner L, van Mechelen W. Predicting older adults' maintenance in exercise participation using an integrated social psychological model. Health Educ Res. 2006 Feb;21(1):1-14. doi: 10.1093/her/cyh037. Epub 2005 Jun 24. PMID 15980075
- [Result] Campbell AJ, Robertson MC, Gardner MM, Norton RN, Tilyard MW, Buchner DM. Randomised controlled trial of a general practice programme of home based exercise to prevent falls in elderly women. BMJ. 1997 Oct 25;315(7115):1065-9. doi: 10.1136/bmj.315.7115.1065. PMID 9366737
- [Result] Cederbom S, Arkkukangas M. Impact of the fall prevention Otago Exercise Programme on pain among community-dwelling older adults: a short- and long-term follow-up study. Clin Interv Aging. 2019 Apr 26;14:721-726. doi: 10.2147/CIA.S200188. eCollection 2019. PMID 31118594
- [Result] Shiri R, Coggon D, Falah-Hassani K. Exercise for the Prevention of Low Back Pain: Systematic Review and Meta-Analysis of Controlled Trials. Am J Epidemiol. 2018 May 1;187(5):1093-1101. doi: 10.1093/aje/kwx337. PMID 29053873
- [Result] O'Sullivan PB, Phyty GD, Twomey LT, Allison GT. Evaluation of specific stabilizing exercise in the treatment of chronic low back pain with radiologic diagnosis of spondylolysis or spondylolisthesis. Spine (Phila Pa 1976). 1997 Dec 15;22(24):2959-67. doi: 10.1097/00007632-199712150-00020. PMID 9431633
- [Result] Bystrom MG, Rasmussen-Barr E, Grooten WJ. Motor control exercises reduces pain and disability in chronic and recurrent low back pain: a meta-analysis. Spine (Phila Pa 1976). 2013 Mar 15;38(6):E350-8. doi: 10.1097/BRS.0b013e31828435fb. PMID 23492976
- [Result] Gross A, Kay TM, Paquin JP, Blanchette S, Lalonde P, Christie T, Dupont G, Graham N, Burnie SJ, Gelley G, Goldsmith CH, Forget M, Hoving JL, Bronfort G, Santaguida PL; Cervical Overview Group. Exercises for mechanical neck disorders. Cochrane Database Syst Rev. 2015 Jan 28;1(1):CD004250. doi: 10.1002/14651858.CD004250.pub5. PMID 25629215
- [Result] Liao CD, Tsauo JY, Huang SW, Ku JW, Hsiao DJ, Liou TH. Effects of elastic band exercise on lean mass and physical capacity in older women with sarcopenic obesity: A randomized controlled trial. Sci Rep. 2018 Feb 2;8(1):2317. doi: 10.1038/s41598-018-20677-7. PMID 29396436